CLINICAL TRIAL: NCT02873936
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter, Phase 3 Study to Assess the Efficacy and Safety of Filgotinib Administered for 24 Weeks in Combination With Conventional Synthetic Disease-modifying Anti-rheumatic Drug(s) (csDMARDs) to Subjects With Moderately to Severely Active Rheumatoid Arthritis Who Have an Inadequate Response to Biologic DMARD(s) Treatment
Brief Title: Filgotinib Versus Placebo in Adults With Active Rheumatoid Arthritis (RA) Who Have an Inadequate Response to Biologic Disease-modifying Anti-rheumatic Drug(s) (DMARDs) Treatment
Acronym: FINCH 2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Collaborators: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-417-0302; 2016-000569-21 (EudraCT Number)
Record Dates: First submitted 2016-08-17; First posted 2016-08-22 (Estimated); Results first posted 2021-01-15 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-04

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — GLPG0634

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Filgotinib 200 mg (Experimental): Filgotinib 200 mg + placebo to match filgotinib 100 mg + stable dose of permitted csDMARD(s)
  Interventions: Drug: Filgotinib; Drug: Placebo to match filgotinib; Drug: csDMARDs
- Filgotinib 100 mg (Experimental): Filgotinib 100 mg + placebo to match filgotinib 200 mg + stable dose of permitted csDMARD(s)
  Interventions: Drug: Filgotinib; Drug: Placebo to match filgotinib; Drug: csDMARDs
- Placebo (Placebo Comparator): Placebo to match filgotinib 200 mg + placebo to match filgotinib 100 mg + stable dose of permitted csDMARD(s)
  Interventions: Drug: Placebo to match filgotinib; Drug: csDMARDs

INTERVENTIONS:
Drug: Filgotinib — Tablet(s) administered orally once daily
  Other Names: GS-6034
  Arms: Filgotinib 100 mg; Filgotinib 200 mg
Drug: Placebo to match filgotinib — Tablet(s) administered orally once daily
Drug: csDMARDs — csDMARDs may include one or two of the following: methotrexate (MTX), hydroxychloroquine or chloroquine, sulfasalazine, and/or leflunomide (combination of leflunomide and MTX is not allowed)

SUMMARY:
The primary objective of this study is to evaluate the effects of filgotinib versus placebo for the treatment of signs and symptoms of rheumatoid arthritis (RA) as measured by the percentage of participants achieving an American College of Rheumatology 20% improvement response (ACR20) at Week 12.

ELIGIBILITY:
Key Inclusion Criteria:

* Have a diagnosis of RA (2010 American College of Rheumatology [ACR]/European League Against Rheumatism [EULAR] criteria for RA), and are ACR functional class I-III.
* Have ≥ 6 swollen joints (from a swollen joint count based on 66 joints [SJC66]) and ≥6 tender joints (from a tender joint count based on 68 joints [TJC68]) at screening and Day 1
* Ongoing treatment with a stable prescription of 1 or 2 csDMARDs
* Have received at least one biologic disease modifying antirheumatic drug (bDMARD) for the treatment of RA to which they have had an inadequate response or intolerance

Key Exclusion Criteria:

* Previous treatment with any janus kinase (JAK) inhibitor

NOTE: Other protocol Inclusion/ Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 449 (Actual)
Dates: Start 2016-07-27 (Actual); Primary Completion 2018-03-20 (Actual); Study Completion 2018-06-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (104):
- United States (55):
  - Huntsville, Alabama
  - Gilbert, Arizona
  - Covina, California
  - Hemet, California
  - La Jolla, California
  - Palm Desert, California
  - Palo Alto, California
  - Riverside, California
  - Upland, California
  - Victorville, California
  - Whittier, California
  - Aventura, Florida
  - DeBary, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Orlando, Florida
  - Plantation, Florida
  - Port Richey, Florida
  - Decatur, Georgia
  - Kansas City, Kansas
  - Wichita, Kansas
  - Elizabethtown, Kentucky
  - Lexington, Kentucky
  - Cumberland, Maryland
  - Frederick, Maryland
  - Worcester, Massachusetts
  - Detroit, Michigan
  - Saint Clair Shores, Michigan
  - Hattiesburg, Mississippi
  - Tupelo, Mississippi
  - St Louis, Missouri
  - Lincoln, Nebraska
  - Lebanon, New Hampshire
  - Freehold, New Jersey
  - Toms River, New Jersey
  - Brooklyn, New York
  - Charlotte, North Carolina
  - Greenville, North Carolina
  - Salisbury, North Carolina
  - Middleburg Heights, Ohio
  - Oklahoma City, Oklahoma
  - Tulsa, Oklahoma
  - Philadelphia, Pennsylvania
  - Wyomissing, Pennsylvania
  - Charleston, South Carolina
  - Columbia, South Carolina
  - Myrtle Beach, South Carolina
  - Orangeburg, South Carolina
  - Memphis, Tennessee
  - Beaumont, Texas
  - Corpus Christi, Texas
  - Mesquite, Texas
  - Plano, Texas
  - San Antonio, Texas
  - Webster, Texas
- Argentina (3):
  - Buenos Aires
  - Caba
  - San Juan
- Victoria Park, Western Australia, Australia
- Belgium (3):
  - Ghent
  - Leuven
  - Merksem
- Montpellier, France
- Germany (3):
  - Berlin
  - Hamburg
  - Ratingen
- Hungary (3):
  - Budapest
  - Gyula
  - Székesfehérvár
- Israel (2):
  - Haifa
  - Ramat Gan
- Japan (15):
  - Hiroshima
  - Izumo
  - Katō
  - Kawagoe
  - Kumamoto
  - Narashino
  - Okayama
  - Sagamihara
  - Sapporo
  - Shinjuku-Ku
  - Takaoka
  - Takasaki
  - Tokorozawa
  - Tokyo
  - Tomigusuku
- Mexico (3):
  - Chihuahua City
  - Distrito Federal
  - Mérida
- Poland (4):
  - Bialystok
  - Poznan
  - Warsaw
  - Wroclaw
- Seoul, South Korea
- Spain (4):
  - Madrid
  - Málaga
  - Sabadell
  - Valencia
- Sankt Gallen, Switzerland
- United Kingdom (5):
  - Doncaster
  - Edinburgh
  - Goodmayes
  - Harlow
  - Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Genovese MC, Kalunian KC, Walker D, Gottenberg JE, De Vlam K, Mozaffarian N, et al. Safety and Efficacy of Filgotinib in a Phase 3 Trial of Patients with Active Rheumatoid Arthritis and Inadequate Response or Intolerance to Biologic Dmards [Abstract No. L06]. ACR/ARHP Annual Meeting; 2018 19-24 October; Chicago, IL, USA.
- [Result] Genovese MC, Kalunian K, Gottenberg JE, Mozaffarian N, Bartok B, Matzkies F, Gao J, Guo Y, Tasset C, Sundy JS, de Vlam K, Walker D, Takeuchi T. Effect of Filgotinib vs Placebo on Clinical Response in Patients With Moderate to Severe Rheumatoid Arthritis Refractory to Disease-Modifying Antirheumatic Drug Therapy: The FINCH 2 Randomized Clinical Trial. JAMA. 2019 Jul 23;322(4):315-325. doi: 10.1001/jama.2019.9055. PMID 31334793
- [Derived] Taylor PC, Downie B, Han L, Hawtin R, Hertz A, Moots RJ, Takeuchi T. Patients with High Baseline Neutrophil-to-Lymphocyte Ratio Exhibit Better Response to Filgotinib as Treatment for Rheumatoid Arthritis. Rheumatol Ther. 2024 Oct;11(5):1383-1392. doi: 10.1007/s40744-024-00695-w. Epub 2024 Jul 10. PMID 38985247
- [Derived] Curtis JR, Emery P, Downie B, Zhong Y, Liu J, Han L, Hawtin RE, Burmester GR. Filgotinib Demonstrates Efficacy in Rheumatoid Arthritis Independent of Smoking Status: Post Hoc Analysis of Phase 3 Trials and Claims-Based Analysis. Rheumatol Ther. 2024 Feb;11(1):177-189. doi: 10.1007/s40744-023-00619-0. Epub 2023 Dec 6. PMID 38057656
- [Derived] Balsa A, Wassenberg S, Tanaka Y, Tournadre A, Orzechowski HD, Rajendran V, Lendl U, Stiers PJ, Watson C, Caporali R, Galloway J, Verschueren P. Effect of Filgotinib on Body Mass Index (BMI) and Effect of Baseline BMI on the Efficacy and Safety of Filgotinib in Rheumatoid Arthritis. Rheumatol Ther. 2023 Dec;10(6):1555-1574. doi: 10.1007/s40744-023-00599-1. Epub 2023 Sep 25. PMID 37747626
- [Derived] Combe B, Besuyen R, Gomez-Centeno A, Matsubara T, Sancho Jimenez JJ, Yin Z, Buch MH. Geographic Analysis of the Safety and Efficacy of Filgotinib in Rheumatoid Arthritis. Rheumatol Ther. 2023 Feb;10(1):35-51. doi: 10.1007/s40744-022-00494-1. Epub 2022 Oct 7. PMID 36205910
- [Derived] Bingham CO 3rd, Walker D, Nash P, Lee SJ, Ye L, Hu H, Khalid JM, Combe B. The impact of filgotinib on patient-reported outcomes and health-related quality of life for patients with active rheumatoid arthritis: a post hoc analysis of Phase 3 studies. Arthritis Res Ther. 2022 Jan 3;24(1):11. doi: 10.1186/s13075-021-02677-7. PMID 34980223
- [Derived] Takeuchi T, Matsubara T, Atsumi T, Amano K, Ishiguro N, Sugiyama E, Yamaoka K, Genovese MC, Kalunian K, Walker D, Gottenberg JE, de Vlam K, Bartok B, Pechonkina A, Kondo A, Gao J, Guo Y, Tasset C, Sundy JS, Tanaka Y. Efficacy and safety of filgotinib in Japanese patients with refractory rheumatoid arthritis: Subgroup analyses of a global phase 3 study (FINCH 2). Mod Rheumatol. 2022 Jan 5;32(1):59-67. doi: 10.1080/14397595.2020.1859675. PMID 33274687

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Australia, Asia, Europe, North America, and South America. The first participant was screened on 27 July 2016. The last study visit occurred on 26 June 2018.
Pre-assignment Details: 688 participants were screened. The enrolled participants continued to receive ongoing therapy with permitted protocol specified Conventional Synthetic Disease-Modifying Anti-Rheumatic Drugs (csDMARDs) (ie, methotrexate (MTX), hydroxychloroquine, sulfasalazine, or leflunomide). MTX was not permitted to be used in combination with leflunomide.
Groups:
- Filgotinib 200 mg: Participants were administered filgotinib 200 mg tablet orally, once daily + placebo to match (PTM) filgotinib 100 mg tablet orally, once daily + stable dose of permitted csDMARDs for median exposure of 24.1 weeks.
- Filgotinib 100 mg: Participants were administered filgotinib 100 mg tablet orally, once daily + PTM filgotinib 200 mg tablet orally, once daily + stable dose of permitted csDMARDs for median exposure of 24 weeks.
- Placebo: Participants were administered PTM filgotinib 200 mg tablet orally, once daily + PTM filgotinib 100 mg tablet orally, once daily + stable dose of permitted csDMARDs for median exposure of 24 weeks.
Period: Overall Study
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Started | 148 | 153 | 148
Completed | 135 | 130 | 116
Not Completed | 13 | 23 | 32
Not completed — Withdrew Consent | 4 | 11 | 20
Not completed — Investigator's Discretion | 3 | 5 | 4
Not completed — Adverse Event | 3 | 5 | 3
Not completed — Protocol Violation | 0 | 1 | 3
Not completed — Lost to Follow-up | 1 | 1 | 1
Not completed — Non-compliance With Study Drug | 1 | 0 | 1
Not completed — Randomized but not Dosed | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo | Total
Number analyzed (Participants) | 147 | 153 | 148 | 448
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.0 (12.5) | 55.0 (12.0) | 56.0 (12.1) | 56.0 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120 | 119 | 121 | 360
  Male | 27 | 34 | 27 | 88
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted = local regulators did not allow collection of race information.
  Participants
    Race: American Indian or Alaska Native | 7 | 9 | 10 | 26
    Race: Asian: Japanese | 12 | 15 | 13 | 40
    Race: Asian: Chinese/Taiwanese/Hong Kong Chinese | 0 | 0 | 0 | 0
    Race: Asian: Vietnamese | 1 | 0 | 0 | 1
    Race: Asian: Korean | 2 | 2 | 1 | 5
    Race: Asian: Other | 0 | 3 | 1 | 4
    Race: Black or African American | 14 | 12 | 21 | 47
    Race: Native Hawaiian or Pacific Islander | 0 | 0 | 0 | 0
    Race: White | 110 | 109 | 97 | 316
    Race: Other | 1 | 3 | 2 | 6
    Race: Not Permitted | 0 | 0 | 3 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted = local regulators did not allow collection of ethnicity information.
  Participants
    Ethnicity: Hispanic or Latino | 26 | 40 | 41 | 107
    Ethnicity: Not Hispanic or Latino | 120 | 112 | 107 | 339
    Ethnicity: Not Permitted | 1 | 1 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 87 | 84 | 84 | 255
  Spain | 4 | 7 | 5 | 16
  Germany | 8 | 4 | 3 | 15
  Belgium | 4 | 3 | 6 | 13
  France | 2 | 2 | 5 | 9
  United Kingdom | 2 | 5 | 2 | 9
  South Korea | 2 | 2 | 1 | 5
  Australia | 1 | 1 | 2 | 4
  Israel | 0 | 1 | 2 | 3
  Switzerland | 1 | 1 | 0 | 2
  Poland | 7 | 5 | 7 | 19
  Hungary | 5 | 7 | 4 | 16
  Mexico | 8 | 13 | 9 | 30
  Argentina | 4 | 3 | 5 | 12
  Japan | 12 | 15 | 13 | 40

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved an American College of Rheumatology (ACR) 20% Improvement (ACR20) Response at Week 12
Description: ACR20 response is achieved when the participant has: ≥20% improvement (reduction) from baseline in tender joint count based on 68 joints (TJC68), swollen joint count based on 66 joints (SJC66) and in at least 3 of the following 5 items: physician's global assessment of disease activity (PGA) and subject's global assessment of disease activity (SGA) assessed using visual analog scale (VAS) on a scale of 0-100 [0 and 100 indicating no disease activity and maximum disease activity]; subject's pain assessment using VAS on a scale of 0-100 [0 and 100 indicating no pain and unbearable pain]; health assessment questionnaire-disability index (HAQ-DI) score contains 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities and scored on a scale of 0-3 [0 and 3 indicating without difficulty and unable to do]; high-sensitivity C-reactive protein (hsCRP). Participants with missing outcomes were set as non-responders.
Time Frame: Week 12
Population: The Full Analysis Set included all randomized participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 147 | 153 | 148
percentage of participants | 66.0 [58.0 to 74.0] | 57.5 [49.4 to 65.7] | 31.1 [23.3 to 38.9]
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 12; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 34.9, 95% CI 2-sided [23.5 to 46.3]
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 12; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 26.4, 95% CI 2-sided [15.0 to 37.9]

2. Secondary Outcome: Change From Baseline in the Health Assessment Questionnaire-Disability Index (HAQ-DI) Score at Week 12
Description: The HAQ-DI score is defined as the average of the scores of eight functional categories (dressing and grooming, arising, eating, walking, hygiene, reach, grip, and other activities), usually completed by the participant. Responses in each functional category are collected as 0-3 [0 (without any difficulty) to 3 (unable to do a task in that area), with or without aids or devices]. The eight category scores are averaged into an overall HAQ-DI score on a scale from 0-3 [0 (no disability) to 3 (completely disabled)] when 6 or more categories are non-missing, total possible score is 3. If more than 2 categories are missing, the HAQ-DI score is set to missing. Negative change from baseline indicates improvement (less disability).
Time Frame: Baseline; Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 147 | 153 | 148
score on a scale
  Baseline | 1.70 (0.656) | 1.64 (0.683) | 1.65 (0.633)
  Change from Baseline at Week 12: number analyzed (Participants) | 137 | 140 | 129
  Change from Baseline at Week 12 | -0.55 (0.590) | -0.48 (0.602) | -0.23 (0.547)
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 12. Least squares (LS)-Mean, 95% confidence interval (CI), and P-value were provided from mixed effects model for repeated measure (MMRM). Missing change scores were not imputed using the MMRM approach assuming an unstructured variance-covariance matrix for the repeated measures; Test type: Superiority; p < 0.001, MMRM — MMRM model included treatment, visit (as categorical), treatment by visit, stratification factors, and baseline value as fixed effects, and participants being the random effect; Least Squares Mean Difference = -0.32, 95% CI 2-sided [-0.45 to -0.19], Standard Error of Mean 0.066
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 12. LS-Mean, 95% CI, and P-value were provided from MMRM. Missing change scores were not imputed using the MMRM approach assuming an unstructured variance-covariance matrix for the repeated measures; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.27, 95% CI 2-sided [-0.40 to -0.14], Standard Error of Mean 0.065

3. Secondary Outcome: Percentage of Participants Who Achieved Disease Activity Score for 28 Joint Count Using C-Reactive Protein [DAS28 (CRP)] ≤ 3.2 at Week 12
Description: The DAS28 score is a measure of the participant's disease activity calculated using the tender joint counts (28 joints), swollen joint counts (28 joints), Patient's Global Assessment of Disease Activity (visual analog scale: 0 = no disease activity to 100 = maximum disease activity), and hsCRP (CRP=hsCRP) for a total possible score of 1 to 9.4. Higher values indicate higher disease activity. Participants with missing outcomes were set as non-responders.
Time Frame: Week 12
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 147 | 153 | 148
percentage of participants | 40.8 [32.5 to 49.1] | 37.3 [29.3 to 45.2] | 15.5 [9.4 to 21.7]
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 12; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 25.3, 95% CI 2-sided [14.7 to 35.8]
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 12; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 21.7, 95% CI 2-sided [11.4 to 32.0]

4. Secondary Outcome: Change From Baseline in 36-Item Short Form Survey (SF-36) Physical Component Summary (PCS) Score at Week 12
Description: The SF-36 is a 36-item, self-reported, generic, comprehensive, and health-related quality of life questionnaire based on 8 health domains in 2 components: physical well-being (physical functioning, role-physical, bodily pain, general health perceptions), mental well-being (vitality, social functioning, role-emotional, and mental health). Each domain is scored by summing the individual items and transforming the scores into a 0 to 100 scale with highest possible score of 100. Higher scores indicate better health status or functioning. Positive change in value indicates improvement and better quality of life.
Time Frame: Baseline; Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 146 | 153 | 148
score on a scale
  Baseline | 30.4 (7.75) | 31.7 (7.76) | 31.1 (8.17)
  Change from Baseline at Week 12: number analyzed (Participants) | 141 | 144 | 133
  Change from Baseline at Week 12 | 7.6 (7.68) | 6.8 (8.22) | 3.6 (8.16)
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 12. LS-Mean, 95% CI, and P-value were provided from MMRM. Missing change scores were not imputed using the MMRM approach assuming an unstructured variance-covariance matrix for the repeated measures; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 4.3, 95% CI 2-sided [2.5 to 6.1], Standard Error of Mean 0.92
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 3.4, 95% CI 2-sided [1.6 to 5.2], Standard Error of Mean 0.92

5. Secondary Outcome: Percentage of Participants Who Achieved DAS28 (CRP) < 2.6 at Week 24
Description: The DAS28 score is a measure of the participant's disease activity calculated using the tender joint counts (28 joints), swollen joint counts (28 joints), Patient's Global Assessment of Disease Activity (visual analog scale: 0 = no disease activity to 100 = maximum disease activity), and hsCRP for a total possible score of 1 to 9.4. Higher values indicate higher disease activity. Participants with missing outcomes were set as non-responders.
Time Frame: Week 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 147 | 153 | 148
percentage of participants | 30.6 [22.8 to 38.4] | 26.1 [18.9 to 33.4] | 12.2 [6.6 to 17.8]
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 24; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 18.5, 95% CI 2-sided [8.6 to 28.3]
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 24; Test type: Superiority; p = 0.003, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 14.0, 95% CI 2-sided [4.6 to 23.4]

6. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy (FACIT)-Fatigue Score at Week 12
Description: FACIT-Fatigue scale is a brief, 13-item, symptom-specific questionnaire that specifically assesses the self-reported severity of fatigue and its impact upon daily activities and functioning in the past 7 days. The FACIT-Fatigue uses 0 (not at all) to 4 (very much) numeric rating scales for a total possible score of 0 to 52. Positive change in value indicates improvement (no or less severity of fatigue).
Time Frame: Baseline; Week 12
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 146 | 152 | 147
score on a scale
  Baseline | 24.2 (11.47) | 23.7 (12.30) | 25.4 (10.89)
  Change from Baseline at Week 12: number analyzed (Participants) | 140 | 143 | 132
  Change from Baseline at Week 12 | 9.6 (11.24) | 8.3 (10.80) | 4.5 (10.37)
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 5.0, 95% CI 2-sided [2.6 to 7.3], Standard Error of Mean 1.19
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.007, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 3.2, 95% CI 2-sided [0.9 to 5.5], Standard Error of Mean 1.18

7. Secondary Outcome: Percentage of Participants Who Achieved ACR 50% Improvement (ACR50) at Weeks 4, 12, and 24
Description: ACR50 response is achieved when the participant has: ≥50% improvement (reduction) from baseline in TJC68, SJC66 and in at least 3 of the following 5 items: PGA and SGA assessed using VAS on a scale of 0-100 [0 and 100 indicating no disease activity and maximum disease activity]; subject's pain assessment using VAS on a scale of 0-100 [0 and 100 indicating no pain and unbearable pain]; HAQ-DI score contains 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities and scored on a scale of 0-3 [0 and 3 indicating without difficulty and unable to do]; hsCRP. Participants with missing outcomes were set as non-responders.
Time Frame: Weeks 4, 12, and 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 147 | 153 | 148
percentage of participants
  Week 4 | 22.4 [15.4 to 29.5] | 21.6 [14.7 to 28.4] | 7.4 [2.9 to 12.0]
  Week 12 | 42.9 [34.5 to 51.2] | 32.0 [24.3 to 39.7] | 14.9 [8.8 to 20.9]
  Week 24 | 45.6 [37.2 to 54.0] | 35.3 [27.4 to 43.2] | 18.9 [12.3 to 25.6]
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 4; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 15.0, 95% CI 2-sided [6.4 to 23.7]
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 4; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 14.1, 95% CI 2-sided [5.7 to 22.6]
Statistical Analysis 3: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 12; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 28.0, 95% CI 2-sided [17.5 to 38.5]
Statistical Analysis 4: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 12; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 17.2, 95% CI 2-sided [7.1 to 27.2]
Statistical Analysis 5: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 24; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 26.7, 95% CI 2-sided [15.8 to 37.6]
Statistical Analysis 6: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 24; Test type: Superiority; p = 0.002, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 16.4, 95% CI 2-sided [5.9 to 26.9]

8. Secondary Outcome: Percentage of Participants Who Achieved ACR 70% Improvement (ACR70) at Weeks 4, 12, and 24
Description: ACR70 response is achieved when the participant has: ≥70% improvement (reduction) from baseline in TJC68, SJC66 and in at least 3 of the following 5 items: PGA and SGA assessed using VAS on a scale of 0-100 [0 and 100 indicating no disease activity and maximum disease activity]; subject's pain assessment using VAS on a scale of 0-100 [0 and 100 indicating no pain and unbearable pain]; HAQ-DI score contains 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities and scored on a scale of 0-3 [0 and 3 indicating without difficulty and unable to do]; hsCRP. Participants with missing outcomes were set as non-responders.
Time Frame: Weeks 4, 12, and 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 147 | 153 | 148
percentage of participants
  Week 4 | 6.1 [1.9 to 10.3] | 8.5 [3.8 to 13.2] | 2.7 [0.0 to 5.7]
  Week 12 | 21.8 [14.8 to 28.8] | 14.4 [8.5 to 20.3] | 6.8 [2.4 to 11.1]
  Week 24 | 32.0 [24.1 to 39.9] | 20.3 [13.6 to 27.0] | 8.1 [3.4 to 12.8]
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 4; Test type: Superiority; p = 0.16, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 3.4, 95% CI 2-sided [-1.9 to 8.8]
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 4; Test type: Superiority; p = 0.039, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 5.8, 95% CI 2-sided [-0.0 to 11.6]
Statistical Analysis 3: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 12; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 15.0, 95% CI 2-sided [6.5 to 23.5]
Statistical Analysis 4: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 12; Test type: Superiority; p = 0.036, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 7.6, 95% CI 2-sided [0.1 to 15.2]
Statistical Analysis 5: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 24; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 23.9, 95% CI 2-sided [14.5 to 33.3]
Statistical Analysis 6: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 24; Test type: Superiority; p = 0.004, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 12.2, 95% CI 2-sided [3.7 to 20.6]

9. Secondary Outcome: Percentage of Participants Who Achieved ACR20 Response at Weeks 4, and 24
Description: ACR20 response is achieved when the participant has: ≥20% improvement (reduction) from baseline in TJC68, SJC66 and in at least 3 of the following 5 items: PGA and SGA assessed using VAS on a scale of 0-100 [0 and 100 indicating no disease activity and maximum disease activity]; subject's pain assessment using VAS on a scale of 0-100 [0 and 100 indicating no pain and unbearable pain]; HAQ-DI score contains 20 questions, 8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities and scored on a scale of 0-3 [0 and 3 indicating without difficulty and unable to do]; hsCRP. Participants with missing outcomes were set as non-responders.
Time Frame: Weeks 4, and 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 147 | 153 | 148
percentage of participants
  Week 4 | 51.7 [43.3 to 60.1] | 44.4 [36.2 to 52.6] | 25.7 [18.3 to 33.1]
  Week 24 | 69.4 [61.6 to 77.2] | 54.9 [46.7 to 63.1] | 34.5 [26.5 to 42.5]
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 4; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 26.0, 95% CI 2-sided [14.6 to 37.4]
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 4; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 18.8, 95% CI 2-sided [7.5 to 30.0]
Statistical Analysis 3: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 24; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 34.9, 95% CI 2-sided [23.6 to 46.3]
Statistical Analysis 4: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 24; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 20.4, 95% CI 2-sided [8.8 to 32.1]

10. Secondary Outcome: Change From Baseline in Individual ACR Component: Tender Joint Count Based on 68 Joints (TJC68) at Weeks 4, 12, and 24
Description: TJC was examined on 68 joints of the fingers, elbows, hips, knees, ankles, and toes distal for pain in response to pressure or passive motion at the study time points. Joint pain was scored as 0 = Absent; 1 = Present for each joint. The overall Tender Joint Count ranged from 0 to 68. A negative change from baseline indicates improvement.
Time Frame: Baseline; Weeks 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: tender joint count
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 146 | 153 | 148
tender joint count
  Baseline | 28.0 (16.1) | 26.0 (15.4) | 27.0 (15.5)
  Change from Baseline at Week 4: number analyzed (Participants) | 145 | 149 | 135
  Change from Baseline at Week 4 | -13.0 (13.5) | -11.0 (11.0) | -8.0 (13.8)
  Change from Baseline at Week 12: number analyzed (Participants) | 136 | 139 | 129
  Change from Baseline at Week 12 | -18.0 (14.1) | -16.0 (11.8) | -12.0 (13.4)
  Change from Baseline at Week 24: number analyzed (Participants) | 122 | 112 | 92
  Change from Baseline at Week 24 | -22.0 (14.2) | -19.0 (13.0) | -17.0 (13.3)
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 4. LS-Mean, 95% CI, and P-value were provided from MMRM. Missing change scores were not imputed using the MMRM approach assuming an unstructured variance-covariance matrix for the repeated measures; Test type: Superiority; p = 0.003, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -4.0, 95% CI 2-sided [-7.0 to -1.0], Standard Error of Mean 1.4
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 4. LS-Mean, 95% CI, and P-value were provided from MMRM. Missing change scores were not imputed using the MMRM approach assuming an unstructured variance-covariance matrix for the repeated measures; Test type: Superiority; p = 0.027, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -3.0, 95% CI 2-sided [-6.0 to -0.0], Standard Error of Mean 1.4
Statistical Analysis 3: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -6.0, 95% CI 2-sided [-8.0 to -3.0], Standard Error of Mean 1.3
Statistical Analysis 4: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -4.0, 95% CI 2-sided [-7.0 to -2.0], Standard Error of Mean 1.3
Statistical Analysis 5: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 24. LS-Mean, 95% CI, and P-value were provided from MMRM. Missing change scores were not imputed using the MMRM approach assuming an unstructured variance-covariance matrix for the repeated measures; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -7.0, 95% CI 2-sided [-10.0 to -4.0], Standard Error of Mean 1.5
Statistical Analysis 6: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 24. LS-Mean, 95% CI, and P-value were provided from MMRM. Missing change scores were not imputed using the MMRM approach assuming an unstructured variance-covariance matrix for the repeated measures; Test type: Superiority; p = 0.006, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -4.0, 95% CI 2-sided [-7.0 to -1.0], Standard Error of Mean 1.5

11. Secondary Outcome: Change From Baseline in Individual ACR Component: Swollen Joint Count Based on 66 Joints (SJC66) at Weeks 4, 12, and 24
Description: The total SJC66 was based on 66 joints (same 68 joints counted in TJC68 minus hips). It was derived as the sum of all "1s" (presence of a joint swelling was scored as "1" and the absence of swelling was scored as "0," provided the joint was not replaced or could not be assessed due to other reasons) thus collected with no penalty considered for the joints not assessed or those which had been replaced. The range for SJC66 is 0 to 66. A negative change from baseline indicates improvement.
Time Frame: Baseline; Weeks 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: swollen joint count
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 146 | 153 | 148
swollen joint count
  Baseline | 18.0 (12.5) | 17.0 (12.4) | 17.0 (9.7)
  Change from Baseline at Week 4: number analyzed (Participants) | 145 | 149 | 135
  Change from Baseline at Week 4 | -10.0 (10.6) | -7.0 (9.2) | -7.0 (8.8)
  Change from Baseline at Week 12: number analyzed (Participants) | 136 | 139 | 129
  Change from Baseline at Week 12 | -12.0 (10.5) | -10.0 (8.6) | -8.0 (8.9)
  Change from Baseline at Week 24: number analyzed (Participants) | 122 | 112 | 92
  Change from Baseline at Week 24 | -14.0 (10.3) | -13.0 (10.0) | -12.0 (8.7)
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.008, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -3.0, 95% CI 2-sided [-5.0 to -1.0], Standard Error of Mean 1.0
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 10, analysis 2]; Test type: Superiority; p = 0.65, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.0, 95% CI 2-sided [-2.0 to 1.0], Standard Error of Mean 1.0
Statistical Analysis 3: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -4.0, 95% CI 2-sided [-5.0 to -2.0], Standard Error of Mean 0.9
Statistical Analysis 4: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.008, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -2.0, 95% CI 2-sided [-4.0 to -1.0], Standard Error of Mean 0.9
Statistical Analysis 5: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 10, analysis 5]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -4.0, 95% CI 2-sided [-5.0 to -2.0], Standard Error of Mean 0.9
Statistical Analysis 6: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 10, analysis 6]; Test type: Superiority; p = 0.039, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -2.0, 95% CI 2-sided [-4.0 to -0.0], Standard Error of Mean 0.9

12. Secondary Outcome: Change From Baseline in Individual ACR Component: Subject's Global Assessment of Disease Activity (SGA) at Weeks 4, 12, and 24
Description: SGA was assessed by the participant using a VAS on a scale of 0 (no disease activity) to 100 (maximum disease activity). A negative change from baseline indicates improvement.
Time Frame: Baseline; Weeks 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 147 | 153 | 148
score on a scale
  Baseline | 68.0 (20.6) | 69.0 (20.2) | 70.0 (18.0)
  Change from Baseline at Week 4: number analyzed (Participants) | 146 | 149 | 138
  Change from Baseline at Week 4 | -21.0 (23.2) | -20.0 (26.1) | -10.0 (22.6)
  Change from Baseline at Week 12: number analyzed (Participants) | 137 | 140 | 130
  Change from Baseline at Week 12 | -31.0 (25.9) | -27.0 (28.4) | -14.0 (26.3)
  Change from Baseline at Week 24: number analyzed (Participants) | 123 | 112 | 92
  Change from Baseline at Week 24 | -38.0 (26.8) | -34.0 (28.1) | -24.0 (28.0)
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -12.0, 95% CI 2-sided [-17.0 to -7.0], Standard Error of Mean 2.7
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 10, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -11.0, 95% CI 2-sided [-16.0 to -5.0], Standard Error of Mean 2.7
Statistical Analysis 3: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -18.0, 95% CI 2-sided [-24.0 to -12.0], Standard Error of Mean 3.0
Statistical Analysis 4: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -13.0, 95% CI 2-sided [-19.0 to -7.0], Standard Error of Mean 3.0
Statistical Analysis 5: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 10, analysis 5]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -18.0, 95% CI 2-sided [-25.0 to -12.0], Standard Error of Mean 3.4
Statistical Analysis 6: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 10, analysis 6]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -13.0, 95% CI 2-sided [-19.0 to -6.0], Standard Error of Mean 3.4

13. Secondary Outcome: Change From Baseline in Individual ACR Component: Physician's Global Assessment of Disease Activity (PGA) at Weeks 4, 12, and 24
Description: PGA was assessed by the physician using a VAS on a scale of 0 (no disease activity) to 3 (maximum disease activity). A negative change from baseline indicates improvement.
Time Frame: Baseline; Weeks 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 147 | 153 | 148
score on a scale
  Baseline | 69.0 (17.6) | 68.0 (18.7) | 66.0 (16.7)
  Change from Baseline at Week 4: number analyzed (Participants) | 145 | 146 | 136
  Change from Baseline at Week 4 | -32.0 (25.2) | -30.0 (24.3) | -19.0 (22.2)
  Change from Baseline at Week 12: number analyzed (Participants) | 132 | 138 | 128
  Change from Baseline at Week 12 | -45.0 (25.2) | -41.0 (26.7) | -28.0 (26.9)
  Change from Baseline at Week 24: number analyzed (Participants) | 122 | 111 | 92
  Change from Baseline at Week 24 | -53.0 (22.7) | -45.0 (23.8) | -41.0 (23.5)
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p < 0.001, Mixed effects model for repeated measure — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -12.0, 95% CI 2-sided [-17.0 to -7.0], Standard Error of Mean 2.6
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 10, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -10.0, 95% CI 2-sided [-15.0 to -5.0], Standard Error of Mean 2.6
Statistical Analysis 3: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -16.0, 95% CI 2-sided [-22.0 to -11.0], Standard Error of Mean 2.8
Statistical Analysis 4: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -13.0, 95% CI 2-sided [-18.0 to -7.0], Standard Error of Mean 2.7
Statistical Analysis 5: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 10, analysis 5]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -13.0, 95% CI 2-sided [-18.0 to -8.0], Standard Error of Mean 2.7
Statistical Analysis 6: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 10, analysis 6]; Test type: Superiority; p = 0.052, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -5.0, 95% CI 2-sided [-11.0 to 0.0], Standard Error of Mean 2.7

14. Secondary Outcome: Change From Baseline in Individual ACR Component: Subject's Pain Assessment at Weeks 4, 12, and 24
Description: The participant assessed their pain severity using a VAS on a scale of 0 (no pain) to 100 (severe pain). A negative change from baseline indicates improvement.
Time Frame: Baseline; Weeks 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 147 | 153 | 148
score on a scale
  Baseline | 66.0 (21.6) | 67.0 (21.7) | 68.0 (19.9)
  Change from Baseline at Week 4: number analyzed (Participants) | 145 | 148 | 137
  Change from Baseline at Week 4 | -22.0 (24.2) | -20.0 (26.3) | -8.0 (22.6)
  Change from Baseline at Week 12: number analyzed (Participants) | 137 | 140 | 129
  Change from Baseline at Week 12 | -30.0 (27.9) | -27.0 (30.9) | -14.0 (27.0)
  Change from Baseline at Week 24: number analyzed (Participants) | 123 | 113 | 92
  Change from Baseline at Week 24 | -37.0 (28.1) | -35.0 (29.1) | -24.0 (28.3)
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -16.0, 95% CI 2-sided [-21.0 to -10.0], Standard Error of Mean 2.7
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 10, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -14.0, 95% CI 2-sided [-19.0 to -8.0], Standard Error of Mean 2.7
Statistical Analysis 3: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -17.0, 95% CI 2-sided [-23.0 to -11.0], Standard Error of Mean 3.1
Statistical Analysis 4: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -13.0, 95% CI 2-sided [-19.0 to -7.0], Standard Error of Mean 3.1
Statistical Analysis 5: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 10, analysis 5]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -16.0, 95% CI 2-sided [-23.0 to -10.0], Standard Error of Mean 3.4
Statistical Analysis 6: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 10, analysis 6]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -12.0, 95% CI 2-sided [-19.0 to -5.0], Standard Error of Mean 3.4

15. Secondary Outcome: Change From Baseline in Individual ACR Component: HAQ-DI at Weeks 4, and 24
Description: The HAQ-DI score is defined as the average of the scores of eight functional categories (dressing and grooming, arising, eating, walking, hygiene, reach, grip, and other activities), usually completed by the participant. Responses in each functional category are collected as 0 (without any difficulty) to 3 (unable to do a task in that area), with or without aids or devices. The eight category scores are averaged into an overall HAQ-DI score on a scale from 0 (no disability) to 3 (completely disabled). A negative change from baseline indicates improvement.
Time Frame: Baseline; Weeks 4, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 147 | 153 | 148
score on a scale
  Baseline | 1.70 (0.656) | 1.64 (0.683) | 1.65 (0.633)
  Change from Baseline at Week 4: number analyzed (Participants) | 145 | 148 | 137
  Change from Baseline at Week 4 | -0.39 (0.493) | -0.32 (0.539) | -0.18 (0.444)
  Change from Baseline at Week 24: number analyzed (Participants) | 123 | 113 | 92
  Change from Baseline at Week 24 | -0.75 (0.620) | -0.60 (0.660) | -0.42 (0.600)
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.22, 95% CI 2-sided [-0.33 to -0.11], Standard Error of Mean 0.055
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 10, analysis 2]; Test type: Superiority; p = 0.006, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.15, 95% CI 2-sided [-0.26 to -0.04], Standard Error of Mean 0.055
Statistical Analysis 3: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 10, analysis 5]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.36, 95% CI 2-sided [-0.51 to -0.21], Standard Error of Mean 0.075
Statistical Analysis 4: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 10, analysis 6]; Test type: Superiority; p = 0.003, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.22, 95% CI 2-sided [-0.37 to -0.08], Standard Error of Mean 0.075

16. Secondary Outcome: Change From Baseline in Individual ACR Component: High-Sensitivity C-Reactive Protein (hsCRP) at Weeks 4, 12, and 24
Time Frame: Baseline; Weeks 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 147 | 153 | 148
mg/L
  Baseline | 17.21 (18.275) | 21.49 (28.206) | 16.42 (18.321)
  Change from Baseline at Week 4: number analyzed (Participants) | 144 | 145 | 132
  Change from Baseline at Week 4 | -9.55 (18.421) | -12.15 (25.502) | 1.04 (13.942)
  Change from Baseline at Week 12: number analyzed (Participants) | 137 | 138 | 129
  Change from Baseline at Week 12 | -11.86 (19.760) | -12.02 (26.226) | 0.57 (15.178)
  Change from Baseline at Week 24: number analyzed (Participants) | 121 | 113 | 88
  Change from Baseline at Week 24 | -10.87 (19.083) | -11.12 (27.766) | -1.50 (15.889)
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -10.51, 95% CI 2-sided [-13.61 to -7.41], Standard Error of Mean 1.578
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 10, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -8.92, 95% CI 2-sided [-12.02 to -5.82], Standard Error of Mean 1.577
Statistical Analysis 3: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -10.94, 95% CI 2-sided [-14.19 to -7.69], Standard Error of Mean 1.652
Statistical Analysis 4: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -8.98, 95% CI 2-sided [-12.22 to -5.73], Standard Error of Mean 1.651
Statistical Analysis 5: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 10, analysis 5]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -9.87, 95% CI 2-sided [-13.73 to -6.00], Standard Error of Mean 1.964
Statistical Analysis 6: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 10, analysis 6]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -6.89, 95% CI 2-sided [-10.80 to -2.98], Standard Error of Mean 1.987

17. Secondary Outcome: Percentage of Participants Who Achieved an Improvement (Decrease) in the HAQ-DI Score ≥ 0.22 at Weeks 4, 12, and 24
Description: The HAQ-DI score is defined as the average of the scores of eight functional categories (dressing and grooming, arising, eating, walking, hygiene, reach, grip, and other activities), usually completed by the participant. Responses in each functional category are collected as 0 (without any difficulty) to 3 (unable to do a task in that area), with or without aids or devices. The eight category scores are averaged into an overall HAQ-DI score on a scale from 0-3 [0 (no disability) to 3 (completely disabled) when 6 or more categories are non-missing, so total possible score is 3. Improvement is defined as reduction in HAQ-DI, (baseline value - postbaseline value) ≥ 0.22. If more than 2 categories are missing, the HAQ-DI score is set to missing. Participants with missing outcomes were set as non-responders.
Time Frame: Weeks 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 147 | 153 | 148
percentage of participants
  Week 4: number analyzed (Participants) | 144 | 148 | 144
  Week 4 | 60.4 [52.1 to 68.8] | 54.7 [46.4 to 63.1] | 40.3 [31.9 to 48.6]
  Week 12: number analyzed (Participants) | 144 | 148 | 144
  Week 12 | 66.7 [58.6 to 74.7] | 66.2 [58.3 to 74.2] | 44.4 [36.0 to 52.9]
  Week 24: number analyzed (Participants) | 144 | 148 | 144
  Week 24 | 68.8 [60.8 to 76.7] | 54.1 [45.7 to 62.4] | 35.4 [27.3 to 43.6]
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 4; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 20.1, 95% CI 2-sided [8.1 to 32.1]
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 4; Test type: Superiority; p = 0.013, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 14.5, 95% CI 2-sided [2.4 to 26.5]
Statistical Analysis 3: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 12; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 22.2, 95% CI 2-sided [10.3 to 34.1]
Statistical Analysis 4: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 12; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 21.8, 95% CI 2-sided [10.0 to 33.6]
Statistical Analysis 5: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 24; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 33.3, 95% CI 2-sided [21.8 to 44.9]
Statistical Analysis 6: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 24; Test type: Superiority; p = 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 18.6, 95% CI 2-sided [6.8 to 30.5]

18. Secondary Outcome: Change From Baseline in DAS28 (CRP) at Weeks 4, 12, and 24
Description: The DAS28 score is a measure of the participant's disease activity calculated using the tender joint counts (28 joints), swollen joint counts (28 joints), SGA (VAS: 0 = no disease activity to 100 = maximum disease activity), and hsCRP for a total possible score of 1 to 9.4. Higher values indicate higher disease activity. A negative change from baseline indicates improvement.
Time Frame: Baseline; Weeks 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 147 | 153 | 148
score on a scale
  Baseline | 5.9 (1.03) | 5.9 (0.98) | 5.9 (0.86)
  Change from Baseline at Week 4: number analyzed (Participants) | 144 | 145 | 129
  Change from Baseline at Week 4 | -1.7 (1.16) | -1.5 (1.14) | -0.9 (1.14)
  Change from Baseline at Week 12: number analyzed (Participants) | 136 | 137 | 128
  Change from Baseline at Week 12 | -2.4 (1.32) | -2.3 (1.38) | -1.3 (1.33)
  Change from Baseline at Week 24: number analyzed (Participants) | 121 | 111 | 88
  Change from Baseline at Week 24 | -2.9 (1.29) | -2.6 (1.32) | -2.1 (1.28)
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.9, 95% CI 2-sided [-1.1 to -0.6], Standard Error of Mean 0.13
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 10, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.7, 95% CI 2-sided [-0.9 to -0.4], Standard Error of Mean 0.13
Statistical Analysis 3: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -1.2, 95% CI 2-sided [-1.5 to -0.9], Standard Error of Mean 0.15
Statistical Analysis 4: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -1.0, 95% CI 2-sided [-1.3 to -0.7], Standard Error of Mean 0.15
Statistical Analysis 5: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 10, analysis 5]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -1.1, 95% CI 2-sided [-1.5 to -0.8], Standard Error of Mean 0.17
Statistical Analysis 6: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 10, analysis 6]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -0.7, 95% CI 2-sided [-1.1 to -0.4], Standard Error of Mean 0.17

19. Secondary Outcome: Percentage of Participants Who Achieved DAS28 (CRP) ≤ 3.2 at Weeks 4, and 24
Description: The DAS28 score is a measure of the participant's disease activity calculated using the tender joint counts (28 joints), swollen joint counts (28 joints), SGA (VAS: 0 = no disease activity to 100 = maximum disease activity), and hsCRP for a total possible score of 1 to 9.4. Higher values indicate higher disease activity. Participants with missing outcomes were set as non-responders.
Time Frame: Weeks 4, and 24
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 147 | 153 | 148
percentage of participants
  Week 4 | 21.8 [14.8 to 28.8] | 22.2 [15.3 to 29.1] | 9.5 [4.4 to 14.5]
  Week 24 | 48.3 [39.9 to 56.7] | 37.9 [29.9 to 45.9] | 20.9 [14.1 to 27.8]
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 4; Test type: Superiority; p = 0.004, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 12.3, 95% CI 2-sided [3.5 to 21.2]
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 4; Test type: Superiority; p = 0.003, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 12.8, 95% CI 2-sided [4.0 to 21.5]
Statistical Analysis 3: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 24; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 27.4, 95% CI 2-sided [16.3 to 38.4]
Statistical Analysis 4: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 24; Test type: Superiority; p = 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 17.0, 95% CI 2-sided [6.2 to 27.7]

20. Secondary Outcome: Percentage of Participants Who Achieved DAS28 (CRP) < 2.6 at Weeks 4, and 12
Description: as for outcome 19
Time Frame: Weeks 4, and 12
Population: Participants in the Full Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 147 | 153 | 148
percentage of participants
  Week 4 | 10.2 [5.0 to 15.4] | 11.8 [6.3 to 17.2] | 2.7 [0.0 to 5.7]
  Week 12 | 22.4 [15.4 to 29.5] | 25.5 [18.3 to 32.7] | 8.1 [3.4 to 12.8]
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 4; Test type: Superiority; p = 0.012, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 7.5, 95% CI 2-sided [1.3 to 13.7]
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 4; Test type: Superiority; p = 0.006, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 9.1, 95% CI 2-sided [2.7 to 15.5]
Statistical Analysis 3: Comparison: Filgotinib 200 mg vs Placebo; Filgotinib 200 mg vs Placebo at Week 12; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 14.3, 95% CI 2-sided [5.6 to 23.1]
Statistical Analysis 4: Comparison: Filgotinib 100 mg vs Placebo; Filgotinib 100 mg vs Placebo at Week 12; Test type: Superiority; p < 0.001, Regression, Logistic — P-value was calculated from the logistic regression with treatment groups and stratification factors in the model; Difference in Response Rates = 17.4, 95% CI 2-sided [8.5 to 26.2]

21. Secondary Outcome: American College of Rheumatology N Percent Improvement (ACR-N) at Weeks 4, 12, and 24
Description: ACR-N is defined as the smallest percentage improvement from baseline in swollen joints, tender joints and the median of the following 5 items (PGA, SGA, subject's pain assessment, HAQ-DI and hsCRP). It has a range between 0 and 100%. PGA and SGA assessed using VAS on a scale of 0-100 [0 and 100 indicating no disease activity and maximum disease activity]; subject's pain assessment using VAS on a scale of 0-100 [0 and 100 indicating no pain and unbearable pain]; HAQ-DI score contains 20 questions,8 components: dressing/grooming, arising, eating, walking, hygiene, reach, grip and activities and scored on a scale of 0-3 [0 and 3 indicating without difficulty and unable to do]. If this calculation results in a negative value, then the ACR-N is set to 0. The ACR-N value indicates an improvement of N%, with higher numbers indicating greater improvement.
Time Frame: Weeks 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percent improvement
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 147 | 153 | 148
percent improvement
  Week 4: number analyzed (Participants) | 139 | 141 | 125
  Week 4 | 26.9 (24.58) | 25.8 (27.09) | 13.7 (19.42)
  Week 12: number analyzed (Participants) | 128 | 135 | 123
  Week 12 | 43.4 (29.26) | 37.1 (30.29) | 19.7 (25.44)
  Week 24: number analyzed (Participants) | 117 | 109 | 86
  Week 24 | 53.5 (27.52) | 45.5 (32.16) | 31.9 (29.52)

22. Secondary Outcome: Number of Participants With European League Against Rheumatism (EULAR) Response at Weeks 4, 12, and 24
Description: Good Response: DAS28(CRP) at visit ≤3.2 and improvement from baseline >1.2.
  Moderate Response: DAS28(CRP) at visit ≤3.2 and improvement from baseline >0.6 and ≤1.2; DAS28(CRP) at visit >3.2 and ≤5.1 and improvement from baseline >0.6; DAS 28(CRP) at visit >5.1 and improvement from baseline >1.2.
  No Response: DAS28(CRP) at visit ≤5.1 and improvement from baseline ≤0.6; DAS 28(CRP) >5.1 at visit and improvement from baseline ≤1.2.
Time Frame: Weeks 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 147 | 153 | 148
Participants
  Week 4: number analyzed (Participants) | 144 | 145 | 129
  Week 4: Good Response | 32 | 34 | 13
  Week 4: Moderate Response | 74 | 65 | 53
  Week 4: No Response | 38 | 46 | 63
  Week 12: number analyzed (Participants) | 136 | 137 | 128
  Week 12: Good Response | 58 | 56 | 23
  Week 12: Moderate Response | 65 | 58 | 51
  Week 12: No Response | 13 | 23 | 54
  Week 24: number analyzed (Participants) | 121 | 111 | 88
  Week 24: Good Response | 70 | 58 | 31
  Week 24: Moderate Response | 43 | 47 | 45
  Week 24: No Response | 8 | 6 | 12

23. Secondary Outcome: Change From Baseline in Clinical Disease Activity Index (CDAI) at Weeks 4, 12, and 24
Description: CDAI is calculated using formula: CDAI = TJC based on 28 joints (TJC28) + SJC based on 28 joints (SJC28) + SGA + PGA. PGA and SGA are assessed using a VAS on a scale of 0-10 [0 and 10 indicating no disease activity and maximum disease activity]. CDAI can range from 0 to 76, with higher score indicating more severe disease activity status. A negative change from baseline indicates improvement.
Time Frame: Baseline; Weeks 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 147 | 153 | 148
score on a scale
  Baseline | 41.7 (14.23) | 40.4 (13.23) | 41.4 (12.00)
  Change from Baseline at Week 4: number analyzed (Participants) | 145 | 146 | 135
  Change from Baseline at Week 4 | -19.1 (13.06) | -16.8 (12.95) | -12.8 (13.71)
  Change from Baseline at Week 12: number analyzed (Participants) | 132 | 137 | 128
  Change from Baseline at Week 12 | -26.2 (15.04) | -23.8 (14.33) | -17.3 (15.22)
  Change from Baseline at Week 24: number analyzed (Participants) | 122 | 110 | 92
  Change from Baseline at Week 24 | -30.9 (13.77) | -27.8 (13.54) | -25.4 (14.40)
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -7.1, 95% CI 2-sided [-10.0 to -4.2], Standard Error of Mean 1.47
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 10, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -5.0, 95% CI 2-sided [-7.9 to -2.2], Standard Error of Mean 1.46
Statistical Analysis 3: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -9.5, 95% CI 2-sided [-12.6 to -6.5], Standard Error of Mean 1.56
Statistical Analysis 4: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -7.6, 95% CI 2-sided [-10.6 to -4.5], Standard Error of Mean 1.55
Statistical Analysis 5: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 10, analysis 5]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -8.7, 95% CI 2-sided [-11.9 to -5.5], Standard Error of Mean 1.64
Statistical Analysis 6: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 10, analysis 6]; Test type: Superiority; p = 0.003, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -4.9, 95% CI 2-sided [-8.2 to -1.6], Standard Error of Mean 1.66

24. Secondary Outcome: Change From Baseline in Simplified Disease Activity Index (SDAI) at Weeks 4, 12, and 24
Description: SDAI is a composite measure that sums the TJC28, SJC28, SGA, PGA, and the hsCRP (in mg/dL). PGA and SGA assessed using VAS on a scale of 0-10 [0 and 10 indicating no disease activity and maximum disease activity]. Higher score indicates more severe disease activity status and total possible score is 0 to 86. A negative change from baseline indicates improvement.
Time Frame: Baseline; Weeks 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 147 | 153 | 148
score on a scale
  Baseline | 43.4 (14.64) | 42.6 (14.16) | 43.0 (12.33)
  Change from Baseline at Week 4: number analyzed (Participants) | 143 | 143 | 129
  Change from Baseline at Week 4 | -20.1 (13.73) | -18.1 (13.19) | -12.9 (14.01)
  Change from Baseline at Week 12: number analyzed (Participants) | 131 | 135 | 127
  Change from Baseline at Week 12 | -27.6 (15.54) | -24.9 (15.01) | -17.2 (15.52)
  Change from Baseline at Week 24: number analyzed (Participants) | 120 | 110 | 88
  Change from Baseline at Week 24 | -32.1 (14.41) | -28.8 (14.19) | -24.9 (14.84)
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -8.1, 95% CI 2-sided [-11.1 to -5.1], Standard Error of Mean 1.52
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 10, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -5.9, 95% CI 2-sided [-8.9 to -2.9], Standard Error of Mean 1.52
Statistical Analysis 3: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -10.7, 95% CI 2-sided [-13.8 to -7.5], Standard Error of Mean 1.60
Statistical Analysis 4: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -8.7, 95% CI 2-sided [-11.8 to -5.5], Standard Error of Mean 1.59
Statistical Analysis 5: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 10, analysis 5]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -10.1, 95% CI 2-sided [-13.5 to -6.8], Standard Error of Mean 1.70
Statistical Analysis 6: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 10, analysis 6]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = -6.1, 95% CI 2-sided [-9.4 to -2.7], Standard Error of Mean 1.71

25. Secondary Outcome: SF-36 PCS Score at Weeks 4, 12, and 24
Description: The SF-36 is a 36-item, self-reported, generic, comprehensive, and health-related quality of life questionnaire based on 8 health domains in 2 components: physical well-being (physical functioning, role-physical, bodily pain, general health perceptions), mental well-being (vitality, social functioning, role-emotional, and mental health). Each domain is scored by summing the individual items and transforming the scores into a 0 to 100 scale with highest possible score of 100. Higher scores indicate better health status or functioning.
Time Frame: Weeks 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 147 | 153 | 148
score on a scale
  Week 4: number analyzed (Participants) | 147 | 149 | 146
  Week 4 | 35.4 (8.72) | 36.4 (9.29) | 33.7 (8.67)
  Week 12: number analyzed (Participants) | 142 | 144 | 133
  Week 12 | 38.3 (10.14) | 38.6 (9.39) | 35.1 (9.90)
  Week 24: number analyzed (Participants) | 123 | 112 | 92
  Week 24 | 40.4 (9.64) | 40.3 (10.31) | 37.7 (9.09)

26. Secondary Outcome: Change From Baseline in SF-36 PCS Score at Weeks 4, and 24
Description: as for outcome 4
Time Frame: Baseline; Weeks 4, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 146 | 153 | 148
score on a scale
  Baseline | 30.4 (7.75) | 31.7 (7.76) | 31.1 (8.17)
  Change from Baseline at Week 4: number analyzed (Participants) | 146 | 149 | 146
  Change from Baseline at Week 4 | 5.1 (6.34) | 4.5 (6.53) | 2.5 (5.91)
  Change from Baseline at Week 24: number analyzed (Participants) | 122 | 112 | 92
  Change from Baseline at Week 24 | 9.4 (8.23) | 9.0 (8.44) | 6.6 (7.95)
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 2.5, 95% CI 2-sided [1.1 to 3.9], Standard Error of Mean 0.70
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 10, analysis 2]; Test type: Superiority; p = 0.005, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 2.0, 95% CI 2-sided [0.6 to 3.4], Standard Error of Mean 0.70
Statistical Analysis 3: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 10, analysis 5]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 3.9, 95% CI 2-sided [1.9 to 5.9], Standard Error of Mean 1.02
Statistical Analysis 4: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 10, analysis 6]; Test type: Superiority; p = 0.002, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 3.1, 95% CI 2-sided [1.1 to 5.2], Standard Error of Mean 1.03

27. Secondary Outcome: SF-36 Mental Component Summary (MCS) Score at Weeks 4, 12, and 24
Description: as for outcome 25
Time Frame: Weeks 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 147 | 153 | 148
score on a scale
  Week 4: number analyzed (Participants) | 147 | 149 | 146
  Week 4 | 48.0 (11.48) | 47.3 (11.51) | 45.5 (11.11)
  Week 12: number analyzed (Participants) | 142 | 144 | 133
  Week 12 | 50.2 (10.58) | 48.8 (11.02) | 47.9 (11.01)
  Week 24: number analyzed (Participants) | 123 | 112 | 92
  Week 24 | 50.6 (10.35) | 49.5 (10.72) | 49.1 (10.56)

28. Secondary Outcome: Change From Baseline in SF-36 MCS Score at Weeks 4, 12, and 24
Description: as for outcome 4
Time Frame: Baseline; Weeks 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 146 | 153 | 148
score on a scale
  Baseline | 44.5 (11.97) | 44.2 (11.59) | 44.3 (11.32)
  Change from Baseline at Week 4: number analyzed (Participants) | 146 | 149 | 146
  Change from Baseline at Week 4 | 3.5 (9.17) | 3.0 (9.03) | 1.2 (9.34)
  Change from Baseline at Week 12: number analyzed (Participants) | 141 | 144 | 133
  Change from Baseline at Week 12 | 5.3 (10.60) | 4.6 (9.76) | 3.7 (9.17)
  Change from Baseline at Week 24: number analyzed (Participants) | 122 | 112 | 92
  Change from Baseline at Week 24 | 6.5 (12.50) | 4.6 (9.22) | 4.3 (9.44)
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.019, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 2.3, 95% CI 2-sided [0.4 to 4.2], Standard Error of Mean 0.97
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 10, analysis 2]; Test type: Superiority; p = 0.073, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 1.7, 95% CI 2-sided [-0.2 to 3.6], Standard Error of Mean 0.97
Statistical Analysis 3: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.045, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 2.1, 95% CI 2-sided [0.0 to 4.1], Standard Error of Mean 1.03
Statistical Analysis 4: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.32, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 1.0, 95% CI 2-sided [-1.0 to 3.0], Standard Error of Mean 1.02
Statistical Analysis 5: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 10, analysis 5]; Test type: Superiority; p = 0.12, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 1.9, 95% CI 2-sided [-0.5 to 4.2], Standard Error of Mean 1.19
Statistical Analysis 6: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 10, analysis 6]; Test type: Superiority; p = 0.96, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 0.1, 95% CI 2-sided [-2.3 to 2.4], Standard Error of Mean 1.20

29. Secondary Outcome: FACIT-Fatigue Score at Weeks 4, 12, and 24
Description: FACIT-Fatigue scale is a brief, 13-item, symptom-specific questionnaire that specifically assesses the self-reported severity of fatigue and its impact upon daily activities and functioning in the past 7 days. The FACIT-Fatigue uses 0 (not at all) to 4 (very much) numeric rating scales for a total possible score of 0 to 52.
Time Frame: Weeks 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 147 | 153 | 148
score on a scale
  Week 4: number analyzed (Participants) | 145 | 144 | 144
  Week 4 | 30.4 (12.48) | 30.3 (12.30) | 27.9 (11.29)
  Week 12: number analyzed (Participants) | 141 | 143 | 132
  Week 12 | 34.0 (12.08) | 32.1 (13.66) | 30.4 (11.79)
  Week 24: number analyzed (Participants) | 123 | 110 | 90
  Week 24 | 36.3 (11.58) | 34.4 (12.51) | 33.3 (11.26)

30. Secondary Outcome: Change From Baseline in FACIT-Fatigue Score at Weeks 4, and 24
Description: as for outcome 6
Time Frame: Baseline; Weeks 4, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 146 | 152 | 147
score on a scale
  Baseline | 24.2 (11.47) | 23.7 (12.30) | 25.4 (10.89)
  Change from Baseline at Week 4: number analyzed (Participants) | 144 | 144 | 144
  Change from Baseline at Week 4 | 6.2 (10.20) | 6.4 (9.87) | 2.2 (8.92)
  Change from Baseline at Week 24: number analyzed (Participants) | 122 | 110 | 90
  Change from Baseline at Week 24 | 11.6 (11.67) | 9.8 (10.39) | 7.0 (10.23)
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 3.7, 95% CI 2-sided [1.6 to 5.7], Standard Error of Mean 1.05
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 10, analysis 2]; Test type: Superiority; p = 0.002, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 3.3, 95% CI 2-sided [1.2 to 5.4], Standard Error of Mean 1.05
Statistical Analysis 3: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 10, analysis 5]; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 4.6, 95% CI 2-sided [2.1 to 7.1], Standard Error of Mean 1.28
Statistical Analysis 4: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 10, analysis 6]; Test type: Superiority; p = 0.11, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 2.1, 95% CI 2-sided [-0.5 to 4.7], Standard Error of Mean 1.30

31. Secondary Outcome: Number of Participants by European Quality of Life 5 Dimensions (EQ-5D) Health Profile Categories at Weeks 4, 12, and 24
Description: The EQ-5D-5 levels (EQ-5D-5L) is a standardized measure of health status of the participant at the visit (same day) that provides a simple, generic measure of health for clinical and economic appraisal. EQ-5D-5L consists of 2 components: a descriptive system of the participant's health and a rating of his or her current health state on a 0-100 VAS. The descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. Rating gets recorded on a vertical VAS in which the endpoints are labeled best imaginable health state is 100 (on the top) and worst imaginable health state is 0 (on the bottom). Higher scores of EQ VAS indicate better health.
Time Frame: Weeks 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 147 | 153 | 148
Participants
  Mobility: Week 4: number analyzed (Participants) | 145 | 144 | 144
  Mobility: Week 4: No Problems | 34 | 45 | 32
  Mobility: Week 4: Slight Problems | 58 | 49 | 49
  Mobility: Week 4: Moderate Problems | 38 | 33 | 36
  Mobility: Week 4: Severe Problems | 15 | 16 | 25
  Mobility: Week 4: Extreme Problems | 0 | 1 | 2
  Mobility: Week 12: number analyzed (Participants) | 141 | 143 | 132
  Mobility: Week 12: No Problems | 47 | 57 | 38
  Mobility: Week 12: Slight Problems | 55 | 48 | 46
  Mobility: Week 12: Moderate Problems | 25 | 29 | 29
  Mobility: Week 12: Severe Problems | 13 | 9 | 19
  Mobility: Week 12: Extreme Problems | 1 | 0 | 0
  Mobility: Week 24: number analyzed (Participants) | 123 | 110 | 90
  Mobility: Week 24: No Problems | 51 | 38 | 32
  Mobility: Week 24: Slight Problems | 38 | 45 | 29
  Mobility: Week 24: Moderate Problems | 23 | 18 | 24
  Mobility: Week 24: Severe Problems | 11 | 8 | 5
  Mobility: Week 24: Extreme Problems | 0 | 1 | 0
  Self-care: Week 4: number analyzed (Participants) | 145 | 144 | 144
  Self-care: Week 4: No Problems | 67 | 67 | 49
  Self-care: Week 4: Slight Problems | 45 | 43 | 52
  Self-care: Week 4: Moderate Problems | 24 | 27 | 28
  Self-care: Week 4: Severe Problems | 6 | 6 | 11
  Self-care: Week 4: Extreme Problems | 3 | 1 | 4
  Self-care: Week 12: number analyzed (Participants) | 141 | 143 | 132
  Self-care: Week 12: No Problems | 79 | 78 | 56
  Self-care: Week 12: Slight Problems | 38 | 46 | 44
  Self-care: Week 12: Moderate Problems | 16 | 15 | 21
  Self-care: Week 12: Severe Problems | 6 | 4 | 11
  Self-care: Week 12: Extreme Problems | 2 | 0 | 0
  Self-care: Week 24: number analyzed (Participants) | 123 | 110 | 90
  Self-care: Week 24: No Problems | 83 | 58 | 45
  Self-care: Week 24: Slight Problems | 23 | 31 | 31
  Self-care: Week 24: Moderate Problems | 13 | 16 | 10
  Self-care: Week 24: Severe Problems | 4 | 4 | 4
  Self-care: Week 24: Extreme Problems | 0 | 1 | 0
  Usual Activities: Week 4: number analyzed (Participants) | 145 | 144 | 144
  Usual Activities: Week 4: No Problems | 27 | 38 | 22
  Usual Activities: Week 4: Slight Problems | 65 | 50 | 44
  Usual Activities: Week 4: Moderate Problems | 26 | 38 | 49
  Usual Activities: Week 4: Severe Problems | 19 | 12 | 25
  Usual Activities: Week 4: Extreme Problems | 8 | 6 | 4
  Usual Activities: Week 12: number analyzed (Participants) | 141 | 143 | 132
  Usual Activities: Week 12: No Problems | 47 | 51 | 26
  Usual Activities: Week 12: Slight Problems | 54 | 41 | 48
  Usual Activities: Week 12: Moderate Problems | 25 | 37 | 38
  Usual Activities: Week 12: Severe Problems | 15 | 11 | 20
  Usual Activities: Week 12: Extreme Problems | 0 | 3 | 0
  Usual Activities: Week 24: number analyzed (Participants) | 123 | 110 | 90
  Usual Activities: Week 24: No Problems | 51 | 41 | 20
  Usual Activities: Week 24: Slight Problems | 45 | 32 | 41
  Usual Activities: Week 24: Moderate Problems | 18 | 28 | 24
  Usual Activities: Week 24: Severe Problems | 8 | 7 | 4
  Usual Activities: Week 24: Extreme Problems | 1 | 2 | 1
  Pain/Discomfort: Week 4: number analyzed (Participants) | 145 | 144 | 144
  Pain/Discomfort: Week 4: No Problems | 8 | 11 | 3
  Pain/Discomfort: Week 4: Slight Problems | 69 | 57 | 37
  Pain/Discomfort: Week 4: Moderate Problems | 45 | 50 | 62
  Pain/Discomfort: Week 4: Severe Problems | 19 | 22 | 36
  Pain/Discomfort: Week 4: Extreme Problems | 4 | 4 | 6
  Pain/Discomfort: Week 12: number analyzed (Participants) | 141 | 143 | 132
  Pain/Discomfort: Week 12: No Problems | 21 | 16 | 10
  Pain/Discomfort: Week 12: Slight Problems | 68 | 56 | 36
  Pain/Discomfort: Week 12: Moderate Problems | 34 | 56 | 57
  Pain/Discomfort: Week 12: Severe Problems | 17 | 14 | 28
  Pain/Discomfort: Week 12: Extreme Problems | 1 | 1 | 1
  Pain/Discomfort: Week 24: number analyzed (Participants) | 123 | 110 | 90
  Pain/Discomfort: Week 24: No Problems | 18 | 20 | 10
  Pain/Discomfort: Week 24: Slight Problems | 61 | 42 | 32
  Pain/Discomfort: Week 24: Moderate Problems | 31 | 36 | 33
  Pain/Discomfort: Week 24: Severe Problems | 12 | 10 | 14
  Pain/Discomfort: Week 24: Extreme Problems | 1 | 2 | 1
  Anxiety/Depression: Week 4: number analyzed (Participants) | 145 | 144 | 144
  Anxiety/Depression: Week 4: No Problems | 78 | 77 | 60
  Anxiety/Depression: Week 4: Slight Problems | 33 | 41 | 43
  Anxiety/Depression: Week 4: Moderate Problems | 25 | 21 | 34
  Anxiety/Depression: Week 4: Severe Problems | 8 | 4 | 5
  Anxiety/Depression: Week 4: Extreme Problems | 1 | 1 | 2
  Anxiety/Depression: Week 12: number analyzed (Participants) | 141 | 143 | 132
  Anxiety/Depression: Week 12: No Problems | 79 | 84 | 71
  Anxiety/Depression: Week 12: Slight Problems | 33 | 30 | 34
  Anxiety/Depression: Week 12: Moderate Problems | 23 | 26 | 23
  Anxiety/Depression: Week 12: Severe Problems | 5 | 3 | 3
  Anxiety/Depression: Week 12: Extreme Problems | 1 | 0 | 1
  Anxiety/Depression: Week 24: number analyzed (Participants) | 123 | 110 | 90
  Anxiety/Depression: Week 24: No Problems | 70 | 62 | 50
  Anxiety/Depression: Week 24: Slight Problems | 33 | 30 | 19
  Anxiety/Depression: Week 24: Moderate Problems | 16 | 13 | 15
  Anxiety/Depression: Week 24: Severe Problems | 4 | 4 | 6
  Anxiety/Depression: Week 24: Extreme Problems | 0 | 1 | 0

32. Secondary Outcome: EQ-5D Current Health VAS at Weeks 4, 12, and 24
Description: EQ-5D-5L is a standardized measure of health status of the participant at the visit (same day) that provides a simple, generic measure of health for clinical and economic appraisal. Participant rates their current health state on a 0-100 VAS. It gets recorded on a vertical VAS in which the endpoints are labeled best imaginable health state is 100 (on the top) and worst imaginable health state is 0 (on the bottom). Higher scores of EQ VAS indicate better health.
Time Frame: Weeks 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 147 | 153 | 148
score on a scale
  Week 4: number analyzed (Participants) | 145 | 144 | 144
  Week 4 | 59.0 (22.1) | 60.0 (19.8) | 52.0 (24.2)
  Week 12: number analyzed (Participants) | 141 | 143 | 132
  Week 12 | 66.0 (23.2) | 65.0 (22.2) | 58.0 (23.0)
  Week 24: number analyzed (Participants) | 123 | 110 | 90
  Week 24 | 70.0 (21.8) | 69.0 (21.3) | 62.0 (23.0)

33. Secondary Outcome: Change From Baseline in EQ-5D Current Health VAS at Weeks 4, 12, and 24
Description: The EQ-5D-5L is a standardized measure of health status of the participant at the visit (same day) that provides a simple, generic measure of health for clinical and economic appraisal. Participant rates their current health state on a 0-100 VAS. It gets recorded on a vertical VAS in which the endpoints are labeled best imaginable health state is 100 (on the top) and worst imaginable health state is 0 (on the bottom). Higher scores of EQ VAS indicate better health. Positive change indicates improvement (better health).
Time Frame: Baseline; Weeks 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 146 | 152 | 147
score on a scale
  Baseline | 49.0 (24.7) | 46.0 (24.0) | 46.0 (22.4)
  Change from Baseline at Week 4: number analyzed (Participants) | 144 | 144 | 144
  Change from Baseline at Week 4 | 10.0 (27.6) | 14.0 (26.8) | 6.0 (26.0)
  Change from Baseline at Week 12: number analyzed (Participants) | 140 | 143 | 132
  Change from Baseline at Week 12 | 17.0 (30.9) | 19.0 (26.4) | 12.0 (26.5)
  Change from Baseline at Week 24: number analyzed (Participants) | 122 | 110 | 90
  Change from Baseline at Week 24 | 22.0 (30.8) | 25.0 (26.7) | 17.0 (25.4)
Statistical Analysis 1: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 10, analysis 1]; Test type: Superiority; p = 0.009, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 6.0, 95% CI 2-sided [2.0 to 11.0], Standard Error of Mean 2.5
Statistical Analysis 2: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 10, analysis 2]; Test type: Superiority; p = 0.003, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 7.0, 95% CI 2-sided [3.0 to 12.0], Standard Error of Mean 2.5
Statistical Analysis 3: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 4, analysis 1]; Test type: Superiority; p = 0.003, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 8.0, 95% CI 2-sided [3.0 to 13.0], Standard Error of Mean 2.6
Statistical Analysis 4: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p = 0.006, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 7.0, 95% CI 2-sided [2.0 to 12.0], Standard Error of Mean 2.6
Statistical Analysis 5: Comparison: Filgotinib 200 mg vs Placebo; [analysis description as in outcome 10, analysis 5]; Test type: Superiority; p = 0.002, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 9.0, 95% CI 2-sided [3.0 to 15.0], Standard Error of Mean 2.9
Statistical Analysis 6: Comparison: Filgotinib 100 mg vs Placebo; [analysis description as in outcome 10, analysis 6]; Test type: Superiority; p = 0.007, MMRM — [p-value comment as in outcome 2, analysis 1]; Least Squares Mean Difference = 8.0, 95% CI 2-sided [2.0 to 14.0], Standard Error of Mean 2.9

34. Secondary Outcome: Work Productivity and Activity Impairment-Rheumatoid Arthritis (WPAI-RA): Mean Percentage of Work Time Missed (Absenteeism) at Weeks 4, 12, and 24
Description: The WPAI is a questionnaire that measures impairments in work activities in participants with RA which consists of 6 questions: Q1-currently employed; Q2-work time missed due to RA; Q3-work time missed due to other reasons; Q4-hours actually worked; Q5-degree RA affected productivity while working (0-10 VAS, with 0 indicating no effect and 10 indicating RA completely prevented the participant from working); Q6-degree RA affected productivity in regular unpaid activities (0-10 VAS, with 0 indicating no effect and 10 indicating RA completely prevented the participant's daily activities). Outcomes are expressed as impairment percentages: Absenteeism (work time missed) due to RA: 100×{Q2/(Q2+Q4)}. Higher numbers indicate greater impairment and less productivity.
Time Frame: Weeks 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of work time missed
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 147 | 153 | 148
percentage of work time missed
  Week 4: number analyzed (Participants) | 39 | 53 | 46
  Week 4 | 8.8 (21.01) | 18.2 (30.93) | 14.3 (27.52)
  Week 12: number analyzed (Participants) | 38 | 48 | 45
  Week 12 | 5.6 (13.79) | 14.6 (27.13) | 12.1 (24.39)
  Week 24: number analyzed (Participants) | 40 | 38 | 30
  Week 24 | 7.6 (16.37) | 13.8 (26.23) | 8.5 (18.08)

35. Secondary Outcome: WPAI-RA: Mean Percentage of Impairment While Working Due to RA (Presenteeism) at Weeks 4, 12, and 24
Description: The WPAI is a questionnaire that measures impairments in work activities in participants with RA which consists of 6 questions: Q1-currently employed; Q2-work time missed due to RA; Q3-work time missed due to other reasons; Q4-hours actually worked; Q5-degree RA affected productivity while working (0-10 VAS, with 0 indicating no effect and 10 indicating RA completely prevented the participant from working); Q6-degree RA affected productivity in regular unpaid activities (0-10 VAS, with 0 indicating no effect and 10 indicating RA completely prevented the participant's daily activities). Outcomes are expressed as impairment percentages: Presenteeism (impairment while working) due to RA: 100×{Q5/10}. Higher numbers indicate greater impairment and less productivity.
Time Frame: Weeks 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of impairment while working
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 147 | 153 | 148
percentage of impairment while working
  Week 4: number analyzed (Participants) | 38 | 49 | 43
  Week 4 | 27.4 (22.50) | 37.8 (25.43) | 48.6 (29.81)
  Week 12: number analyzed (Participants) | 38 | 46 | 43
  Week 12 | 23.9 (20.99) | 34.8 (27.22) | 44.2 (29.21)
  Week 24: number analyzed (Participants) | 40 | 36 | 30
  Week 24 | 28.0 (27.57) | 25.6 (22.10) | 36.7 (26.95)

36. Secondary Outcome: WPAI-RA: Mean Percentage of Overall Work Productivity Impairment Due to RA at Weeks 4, 12, and 24
Description: The WPAI is a questionnaire that measures impairments in work activities in participants with RA which consists of 6 questions: Q1-currently employed; Q2-work time missed due to RA; Q3-work time missed due to other reasons; Q4-hours actually worked; Q5-degree RA affected productivity while working (0-10 VAS, with 0 indicating no effect and 10 indicating RA completely prevented the participant from working); Q6-degree RA affected productivity in regular unpaid activities (0-10 VAS, with 0 indicating no effect and 10 indicating RA completely prevented the participant's daily activities). Outcomes are expressed as impairment percentages: Work productivity loss (overall work impairment) due to RA: 100×{Q2/(Q2+Q4) + [(1-Q2/(Q2+Q4) × (Q5/10)]}. Higher numbers indicate greater impairment and less productivity.
Time Frame: Weeks 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of overall work productivity
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 147 | 153 | 148
percentage of overall work productivity
  Week 4: number analyzed (Participants) | 38 | 49 | 43
  Week 4 | 30.8 (24.36) | 43.1 (27.82) | 51.3 (30.85)
  Week 12: number analyzed (Participants) | 38 | 46 | 43
  Week 12 | 26.9 (24.20) | 39.5 (29.37) | 46.9 (30.63)
  Week 24: number analyzed (Participants) | 40 | 36 | 30
  Week 24 | 31.7 (29.94) | 31.4 (25.65) | 39.8 (29.49)

37. Secondary Outcome: WPAI-RA: Mean Percentage of Activity Impairment Due to RA at Weeks 4, 12, and 24
Description: The WPAI is a questionnaire that measures impairments in work activities in participants with RA which consists of 6 questions: Q1-currently employed; Q2-work time missed due to RA; Q3-work time missed due to other reasons; Q4-hours actually worked; Q5-degree RA affected productivity while working (0-10 VAS, with 0 indicating no effect and 10 indicating RA completely prevented the participant from working); Q6-degree RA affected productivity in regular unpaid activities (0-10 VAS, with 0 indicating no effect and 10 indicating RA completely prevented the participant's daily activities). Outcomes are expressed as impairment percentages: Activity impairment due to RA: 100×{Q6/10}. If Question 1 (Are you currently employed?) is 'NO', then only the activity impairment score can be determined. Higher numbers indicate greater impairment and less productivity.
Time Frame: Weeks 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of activity impairment
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 147 | 153 | 148
percentage of activity impairment
  Week 4: number analyzed (Participants) | 145 | 144 | 144
  Week 4 | 49.6 (26.56) | 49.9 (27.43) | 60.3 (25.49)
  Week 12: number analyzed (Participants) | 141 | 143 | 132
  Week 12 | 40.3 (26.75) | 45.5 (28.23) | 53.0 (27.26)
  Week 24: number analyzed (Participants) | 123 | 110 | 90
  Week 24 | 33.3 (24.61) | 37.5 (27.00) | 45.7 (25.57)

38. Secondary Outcome: Change From Baseline in WPAI-RA: Mean Percentage of Work Time Missed (Absenteeism) at Weeks 4, 12, and 24
Description: The WPAI is a questionnaire that measures impairments in work activities in participants with RA which consists of 6 questions: Q1-currently employed; Q2-work time missed due to RA; Q3-work time missed due to other reasons; Q4-hours actually worked; Q5-degree RA affected productivity while working (0-10 VAS, with 0 indicating no effect and 10 indicating RA completely prevented the participant from working); Q6-degree RA affected productivity in regular unpaid activities (0-10 VAS, with 0 indicating no effect and 10 indicating RA completely prevented the participant's daily activities). Outcomes are expressed as impairment percentages: Absenteeism (work time missed) due to RA: 100×{Q2/(Q2+Q4)}. Higher numbers indicate greater impairment and less productivity. A negative change from baseline indicates improvement.
Time Frame: Baseline; Weeks 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of work time missed
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 35 | 54 | 48
percentage of work time missed
  Baseline | 11.3 (16.31) | 19.2 (28.57) | 10.8 (25.65)
  Change from Baseline at Week 4: number analyzed (Participants) | 34 | 48 | 43
  Change from Baseline at Week 4 | -4.3 (20.98) | -3.4 (24.57) | 4.0 (20.75)
  Change from Baseline at Week 12: number analyzed (Participants) | 31 | 46 | 40
  Change from Baseline at Week 12 | -3.6 (17.60) | -7.0 (30.93) | 3.8 (18.40)
  Change from Baseline at Week 24: number analyzed (Participants) | 29 | 34 | 25
  Change from Baseline at Week 24 | -4.6 (22.50) | -3.1 (34.28) | 3.7 (25.13)

39. Secondary Outcome: Change From Baseline in WPAI-RA: Mean Percentage of Impairment While Working Due to RA (Presenteeism) at Weeks 4, 12, and 24
Description: The WPAI is a questionnaire that measures impairments in work activities in participants with RA which consists of 6 questions: Q1-currently employed; Q2-work time missed due to RA; Q3-work time missed due to other reasons; Q4-hours actually worked; Q5-degree RA affected productivity while working (0-10 VAS, with 0 indicating no effect and 10 indicating RA completely prevented the participant from working); Q6-degree RA affected productivity in regular unpaid activities (0-10 VAS, with 0 indicating no effect and 10 indicating RA completely prevented the participant's daily activities). Outcomes are expressed as impairment percentages: Presenteeism (impairment while working) due to RA: 100×{Q5/10}. Higher numbers indicate greater impairment and less productivity. A negative change from baseline indicates improvement.
Time Frame: Baseline; Weeks 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of impairment while working
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 35 | 51 | 46
percentage of impairment while working
  Baseline | 46.9 (24.71) | 51.0 (27.95) | 55.7 (26.64)
  Change from Baseline at Week 4: number analyzed (Participants) | 34 | 45 | 40
  Change from Baseline at Week 4 | -19.1 (25.63) | -13.1 (25.75) | -5.3 (25.52)
  Change from Baseline at Week 12: number analyzed (Participants) | 31 | 42 | 38
  Change from Baseline at Week 12 | -20.0 (25.56) | -18.8 (28.64) | -10.8 (20.32)
  Change from Baseline at Week 24: number analyzed (Participants) | 29 | 31 | 25
  Change from Baseline at Week 24 | -18.6 (22.48) | -28.7 (25.26) | -20.0 (31.36)

40. Secondary Outcome: Change From Baseline in WPAI-RA: Mean Percentage of Overall Work Productivity Impairment Due to RA at Weeks 4, 12, and 24
Description: The WPAI is a questionnaire that measures impairments in work activities in participants with RA which consists of 6 questions: Q1-currently employed; Q2-work time missed due to RA; Q3-work time missed due to other reasons; Q4-hours actually worked; Q5-degree RA affected productivity while working (0-10 VAS, with 0 indicating no effect and 10 indicating RA completely prevented the participant from working); Q6-degree RA affected productivity in regular unpaid activities (0-10 VAS, with 0 indicating no effect and 10 indicating RA completely prevented the participant's daily activities). Outcomes are expressed as impairment percentages: Work productivity loss (overall work impairment) due to RA: 100×{Q2/(Q2+Q4) + [(1-Q2/(Q2+Q4) × (Q5/10)]}. Higher numbers indicate greater impairment and less productivity. A negative change from baseline indicates improvement.
Time Frame: Baseline; Weeks 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of overall work productivity
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 35 | 51 | 46
percentage of overall work productivity
  Baseline | 52.0 (24.02) | 55.8 (30.53) | 56.7 (27.60)
  Change from Baseline at Week 4: number analyzed (Participants) | 34 | 45 | 40
  Change from Baseline at Week 4 | -20.9 (28.94) | -12.3 (28.05) | -3.4 (25.48)
  Change from Baseline at Week 12: number analyzed (Participants) | 31 | 42 | 38
  Change from Baseline at Week 12 | -22.8 (29.20) | -19.5 (31.49) | -8.3 (20.16)
  Change from Baseline at Week 24: number analyzed (Participants) | 29 | 31 | 25
  Change from Baseline at Week 24 | -20.5 (26.20) | -26.4 (29.87) | -16.7 (33.28)

41. Secondary Outcome: Change From Baseline in WPAI-RA: Mean Percentage of Activity Impairment Due to RA at Weeks 4, 12, and 24
Description: The WPAI is a questionnaire that measures impairments in work activities in participants with RA which consists of 6 questions: Q1-currently employed; Q2-work time missed due to RA; Q3-work time missed due to other reasons; Q4-hours actually worked; Q5-degree RA affected productivity while working (0-10 VAS, with 0 indicating no effect and 10 indicating RA completely prevented the participant from working); Q6-degree RA affected productivity in regular unpaid activities (0-10 VAS, with 0 indicating no effect and 10 indicating RA completely prevented the participant's daily activities). Outcomes are expressed as impairment percentages: Activity impairment due to RA: 100×{Q6/10}. If Question 1 (Are you currently employed?) is 'NO', then only the activity impairment score can be determined. Higher numbers indicate greater impairment and less productivity. A negative change from baseline indicates improvement.
Time Frame: Baseline; Weeks 4, 12, and 24
Population: Participants in the Full Analysis Set with available data were analyzed.
Measure: Mean (Standard Deviation); unit: percentage of activity impairment
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
Number analyzed (Participants) | 146 | 152 | 147
percentage of activity impairment
  Baseline | 65.6 (22.16) | 64.6 (23.07) | 65.4 (23.33)
  Change from Baseline at Week 4: number analyzed (Participants) | 144 | 144 | 144
  Change from Baseline at Week 4 | -16.0 (24.64) | -14.3 (22.89) | -4.7 (25.06)
  Change from Baseline at Week 12: number analyzed (Participants) | 140 | 143 | 132
  Change from Baseline at Week 12 | -25.0 (26.81) | -19.2 (28.32) | -11.3 (25.75)
  Change from Baseline at Week 24: number analyzed (Participants) | 122 | 110 | 90
  Change from Baseline at Week 24 | -32.5 (27.37) | -27.1 (27.97) | -18.4 (31.23)

ADVERSE EVENTS:
Time Frame: First dose date up to last dose date (Maximum: 29.3 weeks) plus 30 days
Description: The Safety Analysis Set included all participants who received at least 1 dose of study drug.
Arm/Group | Filgotinib 200 mg | Filgotinib 100 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/147 | 0/153 | 0/148
Serious Adverse Events (participants affected / at risk) | 6/147 | 8/153 | 5/148
Other Adverse Events (participants affected / at risk) | 39/147 | 35/153 | 31/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Filgotinib 200 mg (N=147) | Filgotinib 100 mg (N=153) | Placebo (N=148)
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 0 | 0 | 1
Abscess oral (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Gallbladder empyema (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 2
Vulval abscess (Infections and infestations) | 0 | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 1 | 0
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Filgotinib 200 mg (N=147) | Filgotinib 100 mg (N=153) | Placebo (N=148)
Nausea (Gastrointestinal disorders) | 7 | 8 | 5
Bronchitis (Infections and infestations) | 8 | 3 | 8
Nasopharyngitis (Infections and infestations) | 15 | 9 | 7
Upper respiratory tract infection (Infections and infestations) | 8 | 9 | 6
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 | 2 | 8
Headache (Nervous system disorders) | 8 | 9 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol: Amendment 1 (2016-07-05): https://cdn.clinicaltrials.gov/large-docs/36/NCT02873936/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-23): https://cdn.clinicaltrials.gov/large-docs/36/NCT02873936/SAP_001.pdf